CLINICAL TRIAL: NCT05271500
Title: Effect of Laser Acupuncture on Immunological Response and Dyspnea in Post Covid Syndrome Patients
Brief Title: New Modality for Post Covid Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Ibrahim Abdelmohsen Alghitany, teacher at faculty of physical therapy, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003582
Record Dates: First submitted 2022-03-07; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Post Covid Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group(1) (Active Comparator): 40 post covid 19 patients will receive laser acupuncture
  Interventions: Device: laser acupuncture
- group(2) (Placebo Comparator): 40 post covid patients will receive placebo laser acupuncture in which laser will be off
  Interventions: Device: laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — gallium-aluminum arsenide diode laser with a continuous wave and a wavelength of 850nm will be used for laser acupuncture. it will be applied for three times per week for 12 weeks

SUMMARY:
Coronavirus (19) is a pandemic that affects many countries allover the world. Many patients experienced symptoms as dyspnea and fatigue after their recovery from coronavirus . These symptoms appear to occur regardless the severity of the infection. In addition, many studies reported change in the inflammatory status and immunity in post covid patients. laser acupuncture is a painless noninvasive modality that is used in treating many diseases. laser acupuncture appear to have a role in relieving symptoms, altering inflammatory status and boosting immunity in post covid patients.

ELIGIBILITY:
Inclusion Criteria:

* age will be ranged from 30 to 40 years
* patients were diagnosed as covid 19 by polymerase chain reaction test using nasopharyngeal swap
* patients will be negative polymerase chain reaction test (pcr) with symptoms of dyspnea and fatigue.
* patients will be recruited after 2 weeks post the negative pcr
* patients who want to participate and complete the study till the end

Exclusion Criteria:

* patients with photosensitivity
* pacemaker plantation pregnant women
* BMI more than 30kg/m2 infection or inflammation at the site of acupuncture laser malignancy uncontrolled diabetes psychiatric disorders or mental retardation

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
change in the level of CD 3 T cells | after 12 weeks of treatment
  5ml of blood will be drawn and serum will be separated. cd3 level will be measured using BD FACS Canto flow cytometer
change in the level of cd4 T cells | after 12 weeks of treatment
  cd4 will be measured using BD FACS Canto flow cytometer after blood sample will be separated
change in level of interleukin 4 | after 12 weeks of treatment
  BD FACS Canto flow cytometer with BD CBA human th1/th2 cytokine kit will be used
change in level of interleukin 6 | after 12 weeks of treatment
  BD FACS Canto flow cytometer with BD CBA human th1/th2 cytokine kit will be used
change in lymphocyte count | after 12 weeks of treatment
  BD FACS Canto flow cytometer will be used
change in level of dyspnea | after 12 weeks of treatment
  mMRC scale is a five point scale to detect degree of dyspnea while performing physical activity. it is ranged from 0-4

SECONDARY OUTCOMES:
change in fatigability | after 12 weeks of treatment
  chalder fatigue scale is 11 items scale. people of 4 or more are considered meeting the criteria of fatigue

CONTACTS AND LOCATIONS:
Overall Officials: shawky fouad, PHD degree, Principal Investigator — Cairo University; sandra girguis, PHD degree, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No